CLINICAL TRIAL: NCT00749619
Title: Addition of Heparin to Taurolock-TM CLS in HD Patients With TCC Dose it Improve Catheter Patency Problems ?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Purpose: Prevention
Other Study IDs: TAURO 070908
Record Dates: First submitted 2008-09-07; First posted 2008-09-09 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: End Stage Renal Disease; Hemodialysis
Keywords: Tunneled Cuffed Catheter; Catheter Lock Solution; Catheter Related Bacteremia
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Citric Acid; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Other: Catheter Lock Solution Taurolidine and Citrate
- B (Experimental)
  Interventions: Other: Catheter Lock Solution :Taurolidine and Citrate and Heparin
- C (No Intervention)
  Interventions: Other: Catheter Lock Solution : Heparin

INTERVENTIONS:
Other: Catheter Lock Solution Taurolidine and Citrate
  Arms: A
Other: Catheter Lock Solution :Taurolidine and Citrate and Heparin
  Arms: B
Other: Catheter Lock Solution : Heparin
  Arms: C

SUMMARY:
Addition of Heparin to the Catheter Lock Solution (CLS): Taurolock-TM will improve the vascular patency compared to Taurolock-TM alone , in hemodialysis patients with Tunneled Cuffed Catheter(TCC) as vascular access.

DETAILED DESCRIPTION:
Bacteremia and thrombosis are the major complications of TCC used for hemodialysis.Instilation of CLS containing antibiotic-anticoagulant solution in the end of each dialysis session till the next dialysis ,can prevent Catheter related bacteremia (CRB).In previous study in our department, Taurolock-TM decreased the rate of CRB but increased the incidence of catheter malfunction.

The aim of the study is to investigate the influence of of Heparin addition to CLS-Taurolock- TM ( Taurolidine &citrate 4%) in prevention of catheter patency problems in HD patients with TCC, in addition to CRB prevention.

Methods : Patients with newly inserted TCC for HD enrolled and randomized to receive one of three CLS types : group 1- Taurolock-TM, Group 2 - Taurolock-TM and Heparin , Group 3- Heparin .Patients were followed for 6 monthes.

The objective of the study is to investigate the effect of Taurolock TM with heparin on the rate of CRB and vascular patency.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients with new TCC
* Informed Consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel